CLINICAL TRIAL: NCT07101211
Title: Effect of Video-Based Information on Anxiety, Depression, and Stress Before Cystoscopy: A Prospective Randomized Controlled Tria
Brief Title: Video Education to Reduce Anxiety and Depression Before Cystoscopy: A Study in First-Time Patients
Acronym: VIDEOCYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enis Mert Yorulmaz (Other)
Collaborators: Izmir Katip Celebi University (Other)
Responsible Party: Sponsor-Investigator, Enis Mert Yorulmaz, Assistant Professor of Urology, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB0242IKCU
Record Dates: First submitted 2025-06-29; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Depression Anxiety Disorder; Stress, Psychological; Cystoscopy
Keywords: Video-based education; Cystoscopy; Anxiety; Psychological stress; Depression
MeSH Terms: conditions — Anxiety Disorders; Stress, Psychological; Depression

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a parallel design to one of two groups: a control group receiving standard written information about cystoscopy, and an intervention group receiving the same written information plus an educational animation video prior to the procedure. Outcomes were assessed pre- and post-procedure in both groups to compare the effects of video-based education on anxiety, stress, and depression levels.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors who evaluated anxiety, stress, and depression scores using the HADS-A, HADS-D, STAI-TX-I, and BDI were blinded to group allocation to reduce assessment bias. This blinding ensured that the assessors were unaware of whether participants had received video-based education or only written information before cystoscopy. The blinding was implemented according to SPIRIT guidelines for clinical trial design to maintain the integrity of outcome evaluations and reduce potential bias in analyzing the psychological effects of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-Based Education + Standard Written Information (Experimental): Participants in this arm received the standard written informed consent form for cystoscopy along with a Turkish-dubbed educational animation video explaining the cystoscopy procedure. The video was provided via a QR code to allow patients to watch it on their mobile devices while waiting for the procedure. The video covered the procedure steps, sensations to expect, and post-procedure care.
  Interventions: Behavioral: Video-Based Educational Animation; Other: Standard Written Informed Consent
- Standard Written Information Only (Active Comparator): Participants in this arm received only the standard written informed consent form describing the cystoscopy procedure. No video-based educational intervention was provided before the procedure.
  Interventions: Other: Standard Written Informed Consent

INTERVENTIONS:
Behavioral: Video-Based Educational Animation — A short, Turkish-dubbed educational animation video explaining the cystoscopy procedure, including steps of the procedure, expected sensations, and post-procedure care. The video is viewed by patients via QR code on their mobile devices before the cystoscopy to enhance patient understanding and reduce anxiety, stress, and depression.
  Arms: Video-Based Education + Standard Written Information
Other: Standard Written Informed Consent — A standard written informed consent form describing the cystoscopy procedure, including the purpose, steps, possible sensations, and post-procedure care, provided to all participants before the procedure.

SUMMARY:
This study looks at whether watching a short educational video before a cystoscopy can help reduce feelings of anxiety, stress, and depression in patients having the procedure for the first time. Cystoscopy is a test that helps doctors see inside the bladder and urinary tract. It can cause worry or fear, especially for patients who have never had it before. In this study, 180 adult patients were divided into two groups. One group received standard written information about the procedure, and the other group received the same written information plus a short, easy-to-understand animation video that explains what will happen during cystoscopy. The video shows what patients might feel, what the procedure looks like, and what to expect afterward. The study measured how patients felt before and after the procedure to see if the video helped them feel calmer and more prepared. The goal is to find out if using videos before medical procedures can improve the patient experience and reduce stress and anxiety.

DETAILED DESCRIPTION:
This prospective, randomized, controlled clinical trial was designed to evaluate the impact of video-based educational interventions on reducing anxiety, depression, and stress levels in patients undergoing cystoscopy for the first time. Cystoscopy is a diagnostic and therapeutic procedure used to examine the bladder and lower urinary tract and may cause significant anxiety and emotional distress, particularly among patients undergoing the procedure for the first time due to its invasive nature and unfamiliarity. This study was conducted at the Urology Clinic of Izmir Katip Celebi University Ataturk Training and Research Hospital, and included 180 adult patients scheduled for their first cystoscopy between May 15 and June 14, 2025.

Participants were randomized using an odd-even allocation method into two groups: (1) the Video Education Group, which received the standard written informed consent document along with a Turkish-dubbed educational animation video explaining the cystoscopy procedure in a clear and patient-friendly manner, and (2) the Control Group, which received only the standard written informed consent document without the video intervention. The educational animation video used in the study was developed by the European Association of Urology (EAU) and adapted with Turkish narration to improve patient comprehension. The video, approximately three minutes in duration, covered the anatomy of the lower urinary tract, the steps of the cystoscopy procedure, the sensations patients may experience during the procedure, and post-procedure expectations such as transient hematuria and mild discomfort. Patients in the video group watched the animation via their personal mobile devices using a QR code approximately 15-20 minutes prior to the procedure while waiting for cystoscopy.

The primary aim of the study was to determine whether the video-based educational intervention could reduce the short-term psychological distress associated with cystoscopy, with a focus on anxiety reduction as the primary outcome. Secondary aims included evaluating the effects of the intervention on stress and depressive symptoms measured using validated psychological assessment tools. These included the Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A) and Depression Subscale (HADS-D), the State-Trait Anxiety Inventory - State Form (STAI TX-I), and the Beck Depression Inventory (BDI), all of which have validated Turkish versions used to ensure consistency and accuracy in the patient population. Pain perception following the procedure was assessed using the Visual Analog Scale (VAS) as an additional secondary outcome. All measurements were taken immediately before the cystoscopy and within 30 minutes after the procedure to capture the acute psychological response to the intervention and the procedure itself.

Patients were included if they were over 18 years of age, scheduled for their first cystoscopy, and provided written informed consent. Exclusion criteria included a history of previous cystoscopy, active urinary tract infections, cognitive impairment, and the use of psychotropic medications, which could confound the psychological assessments. The cystoscopy procedure was performed using a 22Fr rigid cystoscope with a 30-degree optic, following the administration of 10 mL of 2% lidocaine gel intraurethrally for local anesthesia, ensuring standardization across all procedures. All procedures were conducted by the same experienced urology team in a controlled outpatient clinic environment to maintain procedural consistency and reduce operator-related variability.

Statistical analyses were conducted using Jamovi (version 2.6) and R (version 4.4.0). The normality of continuous data was evaluated using the Shapiro-Wilk test. Depending on the distribution, independent samples t-tests or Mann-Whitney U tests were used to compare differences between groups. A 2x2 repeated measures ANOVA was performed to analyze the effects of time (pre- and post-procedure), group (video vs. control), and the interaction between time and group on psychological outcomes. Subgroup analyses based on patients' education and employment status were conducted using multivariate repeated measures ANOVA with Bonferroni-adjusted post-hoc tests to assess the potential moderating effects of these variables on the intervention's effectiveness. Effect sizes were reported using partial eta squared (η²p) to indicate the magnitude of the observed effects.

A priori power analysis was conducted using G*Power version 3.1, with a medium effect size (Cohen's d = 0.50), an alpha level of 0.05, and a desired power of 0.90, indicating a minimum required sample size of 86 participants per group, which was met by the final enrollment of 180 patients, ensuring the study was sufficiently powered to detect statistically significant differences.

The study adhered to ethical principles in accordance with the Declaration of Helsinki and was approved by the Izmir Katip Celebi University Health Research Ethics Committee (IRB#0242, Date: May 15, 2025). Written informed consent was obtained from all participants prior to enrollment in the study. No external funding influenced the study design, data collection, analysis, or reporting, ensuring the objectivity and independence of the research findings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Undergoing first-time cystoscopy
* Provided written informed consent

Exclusion Criteria:

* History of previous cystoscopy
* Active urinary tract infection
* Cognitive impairment
* Current use of psychotropic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-06-14 (Actual); Study Completion 2025-06-14 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety Levels Assessed by HADS-A Before and After Cystoscopy | Immediately before cystoscopy and within 30 minutes post-procedure
  The Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A) assesses anxiety symptoms in patients while minimizing the influence of physical illness.
  It includes 7 items scored from 0 to 3, with a total score range of 0-21. Scores are interpreted as: 0-7 normal, 8-10 borderline, 11-21 abnormal.
  It avoids somatic symptoms and is widely validated across medical settings. The Turkish version used in this study was validated by Aydemir (1997).
  Due to its brevity and focus on emotional symptoms, HADS-A is suitable for measuring procedural anxiety before and after interventions such as cystoscopy.
  Turkish Validation: Aydemir O. Validity and Reliability of Turkish Version of Hospital Anxiety and Depression Scale. Turkish Journal of Psychiatry. 1997 Apr;8:280-7.
Change in Anxiety Levels Assessed by STAI Form TX-I Before and After Cystoscopy | Immediately before cystoscopy and within 30 minutes post-procedure
  The State-Trait Anxiety Inventory - State Form (STAI Form TX-I) is a 20-item self-report scale measuring temporary, situation-specific anxiety.
  Each item is rated on a 4-point Likert scale, with scores ranging from 20 to 80. Higher scores indicate more severe state anxiety. Some items are reverse scored.
  Typical interpretations: 20-37 (low), 38-44 (moderate), ≥45 (high anxiety).
  The Turkish version was validated by Öner & LeCompte (1983). It is widely used in procedural settings to assess acute stress responses and emotional tension before and after interventions such as cystoscopy.
  Turkish Validation: Öner, Necla, William Ayhan LeCompte. Durumluk Surekli Kaygi Envanteri El Kitabi, Bogazici Universitesi Yayinlari, Istanbul, 1-26. (In Turkish). 1983.

SECONDARY OUTCOMES:
Change in Depression Levels Assessed by HADS-D Before and After Cystoscopy | Immediately before cystoscopy and within 30 minutes post-procedure
  The Hospital Anxiety and Depression Scale - Depression Subscale (HADS-D) is a 7-item scale assessing depressive symptoms in medical patients, minimizing confounding from somatic complaints.
  Each item is scored 0-3, for a total score between 0 and 21. Higher scores indicate more severe depression: 0-7 normal, 8-10 borderline, 11-21 abnormal. The scale excludes physical symptoms like fatigue or appetite loss, making it ideal for use in hospital and outpatient settings.
  The Turkish version used in this study was validated by Aydemir (1997) and is widely applied in clinical research.
  Turkish Validation: Aydemir O. Validity and Reliability of Turkish Version of Hospital Anxiety and Depression Scale. Turkish Journal of Psychiatry. 1997 Apr;8:280-7.
Change in Depression Levels Assessed by Beck Depression Inventory (BDI) Before and After Cystoscopy | Immediately before cystoscopy and within 30 minutes post-procedure
  The Beck Depression Inventory (BDI) is a 21-item self-report scale assessing emotional, cognitive, and somatic symptoms of depression.
  Each item includes four response options scored from 0 to 3, with total scores ranging from 0 to 63. Higher scores indicate more severe depression: 0-13 minimal, 14-19 mild, 20-28 moderate, ≥29 severe.
  The Turkish version used in this study was validated by Tekindal et al. (2021).
  BDI is widely used in clinical research to measure depressive symptom severity and to assess changes in mood before and after medical interventions.
  Turkish Validation: Tekindal M, Tekindal MA. Validity and Reliability of Basic Depression Scale For Turkey. Batı Karadeniz Tıp Dergisi. 2021 Dec 25;5(3):452-63.

OTHER OUTCOMES:
Effect of Patient Education Level on Change in Anxiety Levels Measured by the Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A) Before and After Cystoscopy | Immediately before cystoscopy and within 30 minutes post-procedure
  Moderating Effect of Education Level on Anxiety Reduction Assessed by Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A)
  This outcome will assess whether the patient's education level influences the effectiveness of the video-based educational intervention in reducing anxiety levels before and after cystoscopy.
  Anxiety will be measured using the Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A), validated in Turkish.
  Scores range from 0 to 21, with higher scores indicating greater anxiety.
  Education level will be recorded individually and categorized as:
  Illiterate Primary/Secondary School High School University Graduate Comparisons of pre- and post-procedure HADS-A scores will be performed within and between these groups.
Effect of Patient Education Level on Change in State Anxiety Levels Measured by the State-Trait Anxiety Inventory - State Form (STAI TX-I) Before and After Cystoscopy | Immediately before cystoscopy and within 30 minutes post-procedure
  Moderating Effect of Education Level on Anxiety Reduction Assessed by State-Trait Anxiety Inventory - State Form (STAI TX-I)
  This outcome aims to determine whether education level (as categorized above) modifies the impact of video-based education on state anxiety before and after cystoscopy.
  Anxiety will be measured using the State-Trait Anxiety Inventory - State Form (STAI TX-I), Turkish validated version.
  Scores range from 20 to 80, with higher scores indicating more severe anxiety.
  Education level groups (illiterate, primary/secondary school, high school, university graduate) will be used to explore potential interactions with the intervention effect.

CONTACTS AND LOCATIONS:
Overall Officials: Enis M Yorulmaz, Assist Prof, Principal Investigator — Izmir Katip Celebi University
Locations (1):
- Izmir Katip Celebi University Ataturk Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share individual participant data (IPD) from this study. However, IPD may be considered for sharing upon reasonable request from journal editors or qualified researchers, in compliance with institutional policies and data protection regulations.

REFERENCES:
- [Result] McClintock G, Wong E, Mancuso P, Lalak N, Gassner P, Haghighi K, Rathore P, McAulay L, Jeffery N. Music during flexible cystoscopy for pain and anxiety - a patient-blinded randomised control trial. BJU Int. 2021 Oct;128 Suppl 1:27-32. doi: 10.1111/bju.15527. Epub 2021 Jul 30. PMID 34174137
- [Result] Zhang ZS, Wang XL, Xu CL, Zhang C, Cao Z, Xu WD, Wei RC, Sun YH. Music reduces panic: an initial study of listening to preferred music improves male patient discomfort and anxiety during flexible cystoscopy. J Endourol. 2014 Jun;28(6):739-44. doi: 10.1089/end.2013.0705. Epub 2014 Mar 31. PMID 24548148
- [Result] Gauba A, Ramachandra MN, Saraogi M, Geraghty R, Hameed BMZ, Abumarzouk O, Somani BK. Music reduces patient-reported pain and anxiety and should be routinely offered during flexible cystoscopy: Outcomes of a systematic review. Arab J Urol. 2021 Mar 3;19(4):480-487. doi: 10.1080/2090598X.2021.1894814. eCollection 2021. PMID 34881066
- [Result] Kwon OS, Kwon B, Kim J, Kim BH. Effects of Heating Therapy on Pain, Anxiety, Physiologic Measures, and Satisfaction in Patients Undergoing Cystoscopy. Asian Nurs Res (Korean Soc Nurs Sci). 2022 May;16(2):73-79. doi: 10.1016/j.anr.2022.02.002. Epub 2022 Feb 20. PMID 35196580
- See also: Video animation of the cystoscopy procedure (prepared by EAU). This video was shown to the patients in the intervention group with Turkish dubbing. — https://www.youtube.com/watch?v=0faFfYsaOKs

DOCUMENTS (1):
  • Informed Consent Form (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT07101211/ICF_000.pdf